CLINICAL TRIAL: NCT01207739
Title: Persistent Lyme Empiric Antibiotic Study Europe. A Prospective, Randomised Study Comparing Two Prolonged Oral Antibiotic Strategies After Initial Intravenous Ceftriaxone Therapy for Patients With Symptoms of Proven or Possible Persistent Lyme Disease
Brief Title: Persistent Lyme Empiric Antibiotic Study Europe
Acronym: PLEASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sint Maartenskliniek (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLEASE; NL-27344.091.09 (Other Grant/Funding Number: ZonMW); 2009-010939-40 (EudraCT Number)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Lyme Disease; Borrelia Infection
Keywords: Prolonged antibiotic treatment in Lyme disease; Doxycycline; Clarithromycin; Hydroxychloroquine
MeSH Terms: conditions — Lyme Disease; Borrelia Infections | interventions — Doxycycline; Clarithromycin; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Doxycycline (Active Comparator)
  Interventions: Drug: Doxycycline
- Clarithromycin and hydroxychloroquine (Active Comparator)
  Interventions: Drug: Clarithromycin and hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — After open-label i.v. ceftriaxone 2000 mg qd via a peripheral i.v. catheter: oral Doxycycline 100 mg combined with a placebo b.i.d. for 12 weeks
  Other Names: Doxycycline disper; CASnr 564-25-0 (doxycycline); 17086-28-1 (doxycycline monohydraat)
  Arms: Doxycycline
Drug: Clarithromycin and hydroxychloroquine — After open-label i.v. ceftriaxone 2000 mg qd via a peripheral i.v. catheter: clarithromycin 500 mg combined with hydroxychloroquine 200 mg b.i.d. for 12 weeks
  Other Names: Clarithromycine Mylan, RVG 32619; CASnr 81103-11-9; Hydroxychloroquine; Plaquenil, RVG 00853; CASnr 118-42-3 (hydroxychloroquine); 737-36-4 (hydroxychloroquine sulfate)
  Arms: Clarithromycin and hydroxychloroquine
Drug: Placebo — After open-label i.v. ceftriaxone 2000 mg qd via a peripheral i.v. catheter: 12 weeks' course of double placebo b.i.d.
  Arms: Placebo

SUMMARY:
The purpose of the study is to establish whether prolonged antibiotic treatment of patients diagnosed with proven or presumed PLD (as endorsed by the international ILADS guidelines) leads to better patient outcome than short-term treatment as endorsed by the Dutch CBO guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating females who are 18 years or older.
* Women of child-bearing potential must agree to use contraception methods other than oral contraceptives during the study therapy period, since failure of oral contraceptives due to long-term antibiotic use has been described and doxycycline might be teratogenic.
* Patients with presumed or proven PLD. In this study, clinical suspicion of PLD is defined as complaints of musculoskeletal pain, arthritis or arthralgia, neuralgia or sensory disturbances (such as paresthesias or dysesthesias), neuropsychological or cognitive disorders, and persistent fatigue, that are:

  * temporally related to an episode of erythema migrans or otherwise proven symptomatic Lyme disease (defined as within 4 months after erythema migrans as assessed by a physician, or positive biopsy, PCR, culture, intrathecal B. burgdorferi antibodies), OR
  * accompanied by a positive B. burgdorferi IgG or IgM immunoblot (as defined by strict criteria in line with the European Union Concerted Action on Lyme Borreliosis (EUCALB)), regardless of prior ELISA IgG/IgM screening results.
* Subjects must sign a written informed consent form.

Exclusion Criteria:

* Subjects with a known history of allergy or intolerance to tetracyclines, macrolides, hydroxychloroquine or ceftriaxone.
* Subjects who have had more than 5 days of antimicrobial therapy with activity against B. burgdorferi within the previous 4 weeks.
* Subjects with a presumed diagnosis of neuroborreliosis (CSF pleocytosis or intrathecal antibody production) for which intravenous antimicrobial therapy is required.
* Subjects with a known diagnosis of HIV-seropositivity or other immune disorders. (No HIV serologic testing is required for the study).
* Subjects with positive syphilis serology or signs of other spirochetal diseases.
* Subjects with moderate or severe liver disease defined as alkaline phosphatase, ALAT, or ASAT greater than 3 times upper limit of normal.
* Subjects who are receiving and cannot discontinue cisapride, astemizole, terfenadine, barbiturates, phenytoin, or carbamazepine (The concentrations of these drugs may increase during clarithromycin therapy and/or lead to reduced availability of doxycycline).
* Subjects who are currently enrolled on other investigational drug trials or receiving investigational agents.
* Subjects who have been previously randomized into this study.
* Severe physical or psychiatric co-morbidity that interferes with participation in the study protocol, including previous medical diagnosis of rheumatic conditions, chronic fatigue syndrome or chronic pain conditions as well as insufficient command of the Dutch language.
* Co-morbidity that could (partially) account for the symptoms of the subject (e.g. vitamin B12 deficiency, anemia, hypothyroidism).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Global score 36-item Short-form General Health Survey (SF 36) | Week 14
  Because different operationalizations of the term 'Global score 36-item Short-form General Health Survey (SF 36)' exist, the primary outcome measure is specified here as the 'physical component summary score' (PCS) of the RAND-36 Health Status Inventory (RAND SF-36, Hays 1998), which is similar to the Medical Outcomes Study (MOS) 36-item Short-Form General Health Survey (SF-36). The PCS is also known as the physical health composite score (PHC). This specification has been communicated to the local Ethics Committee on March 1, 2011, and was approved on April 6, 2011.

SECONDARY OUTCOMES:
Subscales 36-item Short-form General Health Survey (SF 36) | weeks 0, 14, 26, 40 and 52
  After the last comprehensive outcome assessment at week 40, patients are surveyed by post-study questionnaires at week 52 (protocol version 3.8; dated July 17, 2009; final Ethics Committee approval April 29, 2010).
Actometer recording during 14 days (objective physical activity) | weeks 0, 14 and 40
Measurements of neuropsychological impairment | weeks 0, 14, 26 and 40
Economic evaluation: Questionaire EQ-5D, health consumption and productivity of labour | weeks 0, 14, 26, 40 and 52
  After the last comprehensive outcome assessment at week 40, patients are surveyed by post-study questionnaires at week 52 (protocol version 3.8; dated July 17, 2009; final Ethics Committee approval April 29, 2010).
Fatigue subscale of Checklist Individual Strength (CIS) | weeks 0, 14, 26, 40 and 52
  After the last comprehensive outcome assessment at week 40, patients are surveyed by post-study questionnaires at week 52 (protocol version 3.8; dated July 17, 2009; final Ethics Committee approval April 29, 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Bart-Jan Kullberg, Prof., M.D., Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Sint Maartenskliniek, Nijmegen

REFERENCES:
- [Background] Berende A, ter Hofstede HJ, Donders AR, van Middendorp H, Kessels RP, Adang EM, Vos FJ, Evers AW, Kullberg BJ. Persistent Lyme Empiric Antibiotic Study Europe (PLEASE)--design of a randomized controlled trial of prolonged antibiotic treatment in patients with persistent symptoms attributed to Lyme borreliosis. BMC Infect Dis. 2014 Oct 16;14:543. doi: 10.1186/s12879-014-0543-y. PMID 25318999
- [Result] Berende A, ter Hofstede HJ, Vos FJ, van Middendorp H, Vogelaar ML, Tromp M, van den Hoogen FH, Donders AR, Evers AW, Kullberg BJ. Randomized Trial of Longer-Term Therapy for Symptoms Attributed to Lyme Disease. N Engl J Med. 2016 Mar 31;374(13):1209-20. doi: 10.1056/NEJMoa1505425. PMID 27028911
- [Derived] van Middendorp H, Berende A, Vos FJ, Ter Hofstede HHM, Kullberg BJ, Evers AWM. Expectancies as predictors of symptom improvement after antimicrobial therapy for persistent symptoms attributed to Lyme disease. Clin Rheumatol. 2021 Oct;40(10):4295-4308. doi: 10.1007/s10067-021-05760-1. Epub 2021 May 24. PMID 34031759
- [Derived] Berende A, Agelink van Rentergem J, Evers AWM, Ter Hofstede HJM, Vos FJ, Kullberg BJ, Kessels RPC. Cognitive impairments in patients with persistent symptoms attributed to Lyme disease. BMC Infect Dis. 2019 Oct 7;19(1):833. doi: 10.1186/s12879-019-4452-y. PMID 31590634
- [Derived] Berende A, Ter Hofstede HJM, Vos FJ, Vogelaar ML, van Middendorp H, Evers AWM, Kessels RPC, Kullberg BJ. Effect of prolonged antibiotic treatment on cognition in patients with Lyme borreliosis. Neurology. 2019 Mar 26;92(13):e1447-e1455. doi: 10.1212/WNL.0000000000007186. Epub 2019 Feb 22. PMID 30796143